CLINICAL TRIAL: NCT05196048
Title: Blood Pressure Sensor of Watch-type Device With ECG Technology
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: ASUSTek Computer INC. (Industry)
Collaborators: China Medical University, Taiwan (Other)
Responsible Party: Sponsor
Other Study IDs: CMUH110-REC2-162
Record Dates: First submitted 2022-01-05; First posted 2022-01-19 (Actual); Last update posted 2022-01-19 (Actual); Status verified 2021-09

CONDITIONS: Blood Pressure
Keywords: AI Algorithm, blood pressure

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- No Intervention: No Intervention
  Interventions: Other: No Intervention

INTERVENTIONS:
Other: No Intervention — No Intervention

SUMMARY:
The ASUS Blood Pressure App "ASUS HealthConnect" is a software-only mobile medical application. It is designed to be compatible with ASUS VivoWatch SP watches and mobile phones. Used together to create, record, store, and display blood pressure information. This application determines the systolic and diastolic blood pressure and pulse rate and provides numerical and historical graphs after calibration with the cuff-type upper arm blood pressure monitor. The above data is only captured when the user is resting.

ELIGIBILITY:
1. Inclusion criteria:

   This plan excludes those under 22 years of age, pregnant, and severe cardiovascular and neurological diseases. It is estimated that about 120 subjects will be admitted and divided into three groups:

   (1.1) The first group-High Range: At least 17 subjects over 22 years old with systolic blood pressure exceeding 140mmHg and diastolic blood pressure exceeding 90mmHg.

   (1.2) The second group-Middle Range: at least 17 subjects over 22 years old with systolic blood pressure ranging from 110mmHg to 140mmHg and diastolic blood pressure ranging from 60mmHg to 90mmHg.

   (1.3) The third group-Low Range: at least 17 subjects over 22 years old with systolic blood pressure lower than 110mmHg and diastolic blood pressure lower than 60mmHg.
2. Exclusion criteria:

(2.1) People younger than 22 years old. (2.2) pregnancy. (2.3) the following conditions:

* Arrhythmia
* Prior heart failure or heart attack
* Peripheral vascular disease or compromised circulation
* Valvular disease (diseases concerning the aortic valve)
* Cardiomyopathy
* Other known cardiovascular disease
* End-stage Renal Disease (ESRD)
* Diabetes
* Neurological disorder (for example, tremors)
* Clotting disorder or you are taking prescribed blood thinners
* Tattoo(s) on the wrist where you will wear the ASUS VivoWatch SP

Min Age: 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: From the preparation before the calibration to the completion of the case acceptance, each person will be tested for about 1 hour, and two research nurses will assist in completing the setting and calibration. In the official measurement, the electronic mercury sphygmomanometer, and ASUS HealthConnect with ASUS VivoWatch SP were used to perform alternate measurements for a total of three comparisons to understand the difference in accuracy between the ASUS HealthConnect, the reference sphygmomanometer.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2021-09-21 (Actual); Primary Completion 2022-05-10 (Estimated); Study Completion 2022-09-20 (Estimated)

PRIMARY OUTCOMES:
Level of accordance between the ASUS HealthConnect App (Blood Pressure Monitor) and the sphygmomanometer | 1 hour per individual
  Excerpted from Regulation 5.2.4.1.2 Data analysis The sphygmomanometer-under-test shall meet the following two criteria.
  a) Criterion 1
  1. The differences of the n individual paired determinations of the sphygmomanometer-under-test and of the observers' readings with the reference sphygmomanometer for all subjects, calculated separately for systolic blood pressure and diastolic blood pressure, shall: i) the mean value of the differences be within or equal to ±5,0 mmHg. ii) the standard deviation no greater than 8,0 mmHg(1,07 kPa). iii) the mean value of the differences and the standard deviation shall be calculated and expressed to at least 0,1 mmHg (0,01 kPa).
  2. The reference blood pressure value shall be the average of the observers' readings with the reference sphygmomanometer preceding and following the sphygmomanometerunder-test determination.

CONTACTS AND LOCATIONS:
Overall Officials: Yeh-Pang Chen, MDPHD, Principal Investigator — China Medical University Hospital
Locations (1):
- China Medical University Hsinchu Hospital, Hsinchu, No. 199, Sec. 1, Xinglong Rd., Zhubei City, Taiwan